CLINICAL TRIAL: NCT05821595
Title: A Phase I, Multi-center, Open-label Study With Dose-escalation and Multiple Expansion Cohorts to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of JYB1907 in Subjects With Advanced Solid Tumors
Brief Title: JYB1907 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JY190701
Record Dates: First submitted 2023-03-20; First posted 2023-04-20 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- JYB1907 Dose 1 (Experimental): Five dose levels of JYB1907 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  The dose of JYB1907 is based on the actual body weight as measured prior to each intravenous administration.
  Interventions: Drug: JYB1907
- JYB1907 Dose 2 (Experimental): Five dose levels of JYB1907 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  The dose of JYB1907 is based on the actual body weight as measured prior to each intravenous administration.
  Interventions: Drug: JYB1907
- JYB1907 Dose 3 (Experimental): Five dose levels of JYB1907 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  The dose of JYB1907 is based on the actual body weight as measured prior to each intravenous administration.
  Interventions: Drug: JYB1907
- JYB1907 Dose 4 (Experimental): Five dose levels of JYB1907 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  The dose of JYB1907 is based on the actual body weight as measured prior to each intravenous administration.
  Interventions: Drug: JYB1907
- JYB1907 Dose 5 (Experimental): Five dose levels of JYB1907 are evaluated in the dose escalation part.In the expansion cohort part, the biologically active dose(s) confirmed in the dose escalation part with one or more dosing regimens will be selected.
  The dose of JYB1907 is based on the actual body weight as measured prior to each intravenous administration.
  Interventions: Drug: JYB1907

INTERVENTIONS:
Drug: JYB1907 — for injection
  Other Names: TGF-β inhibitor

SUMMARY:
A Phase I, Multi-center, Open-label Study with Dose-escalation and Multiple Expansion Cohorts to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of JYB1907 in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
Dose escalation This part is meant to evaluate the safety, tolerability, PK, immunogenicity, preliminary antitumor activity, the MTD and RP2D of JYB1907 in patients with histologically or cytologically confirmed advanced solid tumors.

Expansion cohort The antitumor activity, safety, tolerability, PK and immunogenicity of JYB1907 will be further evaluated in other cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent voluntarily;
2. Age ≥18, male or female;
3. Have at least one evaluable lesion (Dose escalation) or measurable lesion;
4. Expected survival ≥12 weeks；
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;

Exclusion Criteria:

1. Received within 4 weeks before the initial treatment, or scheduled during the study to receive a major surgery, live attenuated vaccines, or any anti-tumor therapy.
2. With severe tumor complications.
3. Pregnant or lactating women, or positive serum pregnancy test;
4. Concurrent participation in another interventional study；
5. With other diseases or clinical abnormalities assessed by the Investigator as ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | until either 28 days after last dose of study drug or initiation of new anticancer therapy, whichever occurs first.
  Adverse events, and changes from baseline in vital signs,etc.

SECONDARY OUTCOMES:
Serum concentrations of JYB1907 | until 28 days after last dose of study drug
  JYB1907 assessed by pre-specified methods, and related pharmacokinetic parameters analysis
Serum concentrations of Immunogenicity Analysis | until 28 days after last dose of study drug
  immunogenicity of JYB1907 assessed by pre-specified methods, and related immunogenic features analysis
Serum concentrations of Preliminary antitumor activity | until 28 days after last dose of study drug
  To evaluate the preliminary antitumor activity of JYB1907 in patients with advanced solid tumors assessed by Recist1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be published or presented at scientific meetings in a timely, objective, and clinically meaningful manner that is consistent with good science, industry and regulator guidance, and the need to protect the intellectual property of the sponsor, regardless of the outcome of the trial. The data generated in this clinical trial are the exclusive property of the sponsor and are confidential. For multicenter studies, the first publication or disclosure of study results shall be a complete, joint multicenter publication or disclosure coordinated by the sponsor. Thereafter, any secondary publications will reference the original publication(s). Authorship will be determined by mutual agreement and all authors must meet the criteria for authorship established by the International Committee of Medical Journal Editors.
Supporting Information: Study Protocol
Time Frame: The study has been completed at all study sites for at least 2 years;
Access Criteria: * The results of the study in their entirety have been publicly disclosed by or with the consent of the sponsor in an abstract, manuscript, or presentation form; or
  * The study has been completed at all study sites for at least 2 years;
  * No such communication, presentation, or publication will include the sponsor's confidential information;
  * Each investigator agrees to submit all manuscripts or congress abstracts and posters/presentations to the sponsor at least 30 days prior to submission. This allows the sponsor to protect confidential information, provide comments based on information from other studies that may not yet be available to the investigator, and ensure scientific and clinical accuracy.